CLINICAL TRIAL: NCT06431685
Title: Phase I Study of Whole Brain Low Dose Radiotherapy Combined With ICI and Intrathecal Chemotherapy for Treatment of Refractory Meningeal Metastasis of Lung Cancer
Brief Title: Safety and Efficacy of Whole Brain LDRT+ICI+Intrathecal Chemotherapy in Refractory Meningeal Metastasis of Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, You Lu, Chair of Department of Thoracic Cancer, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LM-001
Record Dates: First submitted 2024-05-19; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: NSCLC; Low Dose Radiotherapy; PD-1 Inhibitor; Leptomeningeal Metastasis
MeSH Terms: conditions — Meningeal Carcinomatosis | interventions — Radiotherapy; Pemetrexed; sintilimab; Immune Checkpoint Inhibitors; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- whole brain LDRT + ICI + intrathecal chemotherapy (Experimental): The treatment regimen consisted of intrathecal chemotherapy (via lumbar puncture, pemetrexed 30 mg, once per three weeks, 4 cycles in total), PD-1 inhibitor (Sintilimab, via intravenous infusion, once per three weeks, 4 cycles in total)), pemetrexed chemotherapy (via intravenous infusion, once per three weeks, 4 cycles in total) and radiotherapy. Whole brain LDRT will be administered at 3 cohorts with increasing dose fractions: 4 Gy/2f of 2 fraction (administered a daily dose of 2 Gy for two days) in group 1; 4 Gy/2f of 4 fractions (administered a daily dose of 2 Gy for two days, once per three weeks, 2 cycles in total) in group 2; 4 Gy/2f of 8 fractions (administered a daily dose of 2 Gy for two days, once per three weeks, 4 cycles in total) in group 3.
  Interventions: Radiation: Whole Brain Low Dose Radiotherapy; Drug: Pemetrexed; Drug: Sintilimab; Drug: Chemotherapy

INTERVENTIONS:
Radiation: Whole Brain Low Dose Radiotherapy — Whole brain LDRT will be administered at 3 cohorts with increasing dose fractions: Group 1: 4 Gy/2f of one cycle; Group 2: 4 Gy/2f of two cycles (Q3w); Group 3: 4 Gy/2f of three cycles (Q3w). WB-LDRT will be administered in a 4 Gy of 2 fractions over two days, starting from Day 1 in the first cycle (a daily dose of 2 Gy, 4 Gy/2f for one cycle, once per three weeks, at minmum in one cycle and maximum in four cycles in total).
  Other Names: WB-LDRT
Drug: Pemetrexed — Pemetrexed, 30 mg, intrathecal injection, once per three weeks, 4 cycles in total
  Other Names: Intrathecal Chemotherapy
Drug: Sintilimab — PD-1 inhibitor (Sintilimab, dose as recommended in the instruction manual), intravenous infusion, once per three weeks, 4 cycles in total
  Other Names: PD-1 Inhibitor
Drug: Chemotherapy — Pemetrexed at a dose of 500 mg/m^2, intravenous infusion, once per three weeks, 4 cycles in total
  Other Names: One of the standard chemotherapy regimens

SUMMARY:
This phase I study aims to investigate the safety and efficacy of whole brain low dose radiotherapy (WB-LDRT) combined with ICI and intrathecal chemotherapy for treatment of refractory meningeal metastasis of lung cancer.

DETAILED DESCRIPTION:
This exploratory phase I study will be conducted in West China Hospital, Sichuan University. Three cohorts of whole brain low dose radiotherapy (3 patients per cohort) will be enrolled to determine the safety and efficacy of whole brain low dose radiotherapy combined with ICI and intrathecal chemotherapy for treatment of refractory meningeal metastasis of lung cancer.

Subjects who fulfil all the inclusion criteria and none of the exclusion criteria will be enrolled and receive treatment with WB-LDRT at same dose (4 Gy/2f) with diffent cycles (decried as below), PD-1 inhibitor, pemetrexed chemotherapy, and intrathecal pemetrexed every 3 weeks (Q3w) for 4 cycles.

Patients will receive WB-LDRT at 3 cohorts with increasing dose fractions: 4 Gy/2f of one cycle in group 1; 4 Gy/2f of two cycles in group 2; 4 Gy/2f of four cycles in group 3.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old and ≤ 75 years old;
2. Patients with a definite diagnosis of leptomeningeal metastasis by cerebrospinal fluid cytology, or patients with clinical diagnosis combined with tumor history, neuroimaging, clinical manifestations, cerebrospinal fluid examination, etc.;
3. Patients with a clear history of lung carcinoma, including histopathological diagnosis or a combination of cytopathology and imaging, and failure of standard treatment;
4. Efficacy of extracranial lesions SD;
5. Patients with no contraindications to craniocranial radiotherapy were judged by radiotherapy doctors. Subjects who agree to receive immunotherapy, Lumbar puncture, intrathecal chemotherapy, and radiotherapy;
6. Expected survival ≥3 months, PS score ≤3;
7. Agree to provide cerebrospinal fluid, blood and tissue samples for biomarker testing;
8. The main organs function normally, no serious blood, heart, lung, liver, kidney, bone marrow and other functional abnormalities and immune deficiency diseases;
9. One week before enrollment, bone marrow and liver and kidney function met the following criteria:

   ① Hemoglobin ≥80 g/L, neutrophils ≥1.5×10^9/L and platelets ≥70×10^9/L;

   ② Renal function: Cr≤ULN (upper limit of normal) × 1.5, endogenous creatinine clearance (Ccr)≥55 ml/min; Liver function: total bilirubin ≤ULN × 1.5; ALT, AST≤ULN × 2.5; (In case of liver metastasis, total bilirubin should not be higher than 3 times the upper normal limit, and transaminase should not be higher than 5 times the upper normal limit);
10. The fertile women agreed to use contraception during the study period and for 6 months after the study ended; Patients who tested negative for a serum or urine pregnancy test within 7 days prior to joining the study and were not breastfed; Men who agreed to use contraception during the study period and for 6 months after the study ended

Exclusion Criteria:

1. Active autoimmune disease or history of autoimmune diseases;
2. Congenital or acquired immunodeficiency;
3. Uncontrolled cardiac clinical symptoms or diseases;
4. Severe infection or severe comorbidities, such as bleeding peptic ulcer, ileus, heart failure, renal failure, or poorly controlled diabetes;
5. History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
6. Other systemic malignancies within the last 5 years;
7. Allergy to any test drug;
8. Uncontrolled epilepsy, neurological failure, or severe treatment-related neurological impairment, uncontrollable psychosis, and other conditions deemed unsuitable for inclusion by the investigator;
9. Pregnant and lactating women, subjects with reproductive capacity are unwilling to take effective contraceptive measures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Clinical response rate | 48 months
  The RANO proposal for response criteria of leptomeningeal metastasis was used to assess the clinical response in this study.
Incidence of treatment-related adverse events | 48 months
  The incidence of treatment-related adverse events were measured for determing tolerability and safety. Adverse events (AEs) are evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE, version 5.0). Events of grade 3-5 are defined as moderate and severe adverse events.

SECONDARY OUTCOMES:
Neurological progression-free survival (NPFS) | 48 months
  NPFS was defined as time from the start of treatment until neurological progression or death. The neurological progression was determined based on the RANO proposal evaluation criteria which have been established and published on Neuro Oncol.
Overall survival | 48 months
  Survival time was recorded since the date of patient enrollment. All patients were followed up until death or the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: You Lu, MD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cao M, Chen W. Epidemiology of lung cancer in China. Thorac Cancer. 2019 Jan;10(1):3-7. doi: 10.1111/1759-7714.12916. Epub 2018 Nov 28. PMID 30485694
- [Background] Clarke JL, Perez HR, Jacks LM, Panageas KS, Deangelis LM. Leptomeningeal metastases in the MRI era. Neurology. 2010 May 4;74(18):1449-54. doi: 10.1212/WNL.0b013e3181dc1a69. PMID 20439847
- [Background] Remon J, Le Rhun E, Besse B. Leptomeningeal carcinomatosis in non-small cell lung cancer patients: A continuing challenge in the personalized treatment era. Cancer Treat Rev. 2017 Feb;53:128-137. doi: 10.1016/j.ctrv.2016.12.006. Epub 2016 Dec 30. PMID 28110254
- [Background] Gleissner B, Chamberlain MC. Neoplastic meningitis. Lancet Neurol. 2006 May;5(5):443-52. doi: 10.1016/S1474-4422(06)70443-4. PMID 16632315
- [Background] Cheng H, Perez-Soler R. Leptomeningeal metastases in non-small-cell lung cancer. Lancet Oncol. 2018 Jan;19(1):e43-e55. doi: 10.1016/S1470-2045(17)30689-7. PMID 29304362
- [Background] Le Rhun E, Weller M, van den Bent M, Brandsma D, Furtner J, Ruda R, Schadendorf D, Seoane J, Tonn JC, Wesseling P, Wick W, Minniti G, Peters S, Curigliano G, Preusser M; EANO Guidelines Committee and ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Leptomeningeal metastasis from solid tumours: EANO-ESMO Clinical Practice Guideline for diagnosis, treatment and follow-up. ESMO Open. 2023 Oct;8(5):101624. doi: 10.1016/j.esmoop.2023.101624. Epub 2023 Sep 19. PMID 37863528
- [Background] Chamberlain M, Junck L, Brandsma D, Soffietti R, Ruda R, Raizer J, Boogerd W, Taillibert S, Groves MD, Le Rhun E, Walker J, van den Bent M, Wen PY, Jaeckle KA. Leptomeningeal metastases: a RANO proposal for response criteria. Neuro Oncol. 2017 Apr 1;19(4):484-492. doi: 10.1093/neuonc/now183. PMID 28039364
- [Background] Yin K, Li YS, Zheng MM, Jiang BY, Li WF, Yang JJ, Tu HY, Zhou Q, Zhong WZ, Yang XN, Chen HJ, Yan HH, Li LL, Wu YL, Zhang XC. A molecular graded prognostic assessment (molGPA) model specific for estimating survival in lung cancer patients with leptomeningeal metastases. Lung Cancer. 2019 May;131:134-138. doi: 10.1016/j.lungcan.2019.03.015. Epub 2019 Mar 18. PMID 31027690
- [Background] Wang Y, Yang X, Li NJ, Xue JX. Leptomeningeal metastases in non-small cell lung cancer: Diagnosis and treatment. Lung Cancer. 2022 Dec;174:1-13. doi: 10.1016/j.lungcan.2022.09.013. Epub 2022 Oct 1. PMID 36206679
- [Background] Thai K, Prat A. CNS therapeutics: Immune cells break the barriers. Sci Transl Med. 2023 Nov 8;15(721):eadh1150. doi: 10.1126/scitranslmed.adh1150. Epub 2023 Nov 8. PMID 37939159